CLINICAL TRIAL: NCT06080360
Title: The Hopkins Rehabilitation Engagement Rating Scale (HRERS): Cross-cultural Adaptation, Reliability, and Validity of the Turkish Version
Brief Title: The Hopkins Rehabilitation Engagement Rating Scale
Acronym: (HRERS)
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Menekse Safak, Res. Assist., Suleyman Demirel University
Other Study IDs: MS2023/01
Record Dates: First submitted 2023-10-02; First posted 2023-10-12 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Rehabilitation
Keywords: Rehabilitation Engagement; Patient-Reported Outcome Measures; Total Knee Arthroplasty; Hopkins Rehabilitation Engagement Rating Scale; Turkish Version
MeSH Terms: interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient-Reported Outcome Measures — Functional Independence Measurement-FIM, Barthel Index and European Quality of Life-5 Dimensions Questionnaire-EQ-5D, which are self-report based evaluation methods, were applied to patients who received routine treatment and met the inclusion criteria.To determine the patients' level of participation in the treatment, Hopkins was scored by the physiotherapist applying the treatment.

SUMMARY:
Objective: To verify the reliability and validity of the Turkish versions of the Hopkins Rehabilitation Engagement Rating Scale (HRERS) for knee arthroplasty.

Methods: A total of 51 consecutive participants, inpatients of an orthopedic clinic at the university hospital, were recruited between 2021-2022 June. Cronbach's alpha coefficient was used to assess internal consistency. By evaluating the scores of 51 retested patients one week later, the test-retest reliability was determined using the intraclass correlation coefficient (ICC). Pearson's correlation coefficient was used to assess the construct validity.

DETAILED DESCRIPTION:
First of all, permission was obtained from Kortte et al., one of the developers of Hopkins Rehabilitation Engagement Rating Scale (HRERS), to have a Turkish version of HRERS via e-mail before starting the research study. The translation and the cultural adaptation of the Turkish version of the HRERS were accomplished in line with the stages outlined by Beaton et al.. Two independent native Turkish translators performed forward translation. One was a physiotherapist to ensure clinical consistency, and the other was a translator with no medical or clinical background to reveal vague concepts in the original questionnaire. A single consequent Turkish translation was formed from the combination of the two translations The Turkish scale was translated back into English by two English-native speakers who speak Turkish fluently, and the English version of the scale was compared to the original. A group of experts authorized the final version of the document in Turkish, which was backward translation. Translators reviewed the translations and compared certain inconsistencies.

Before the formal questionnaire, the pre-final Turkish version of the questionnaire was used for a pilot test. The Turkish translation was primarily applied to five participants for the detection of unintelligible questions or words. Turkish translation was applied to five participants in order to determine the questions or words that were not understood. We asked the participants the following questions: "Is there a question you don't understand?" "Are there any words you don't like?" Since the participants did not have any problems, no changes were made to the questionnaire, and the final Turkish version of the HRERS (HRERS-T) was provided.

ELIGIBILITY:
Inclusion Criteria:

* Providing hospitalization and rehabilitation follow-up due to knee or hip arthroplasty by Süleyman Demirel University Hospital, Department of Orthopedics and Traumatology,
* Volunteering to participate in the study,
* It means getting a score of 24 or above when the Standardized Mini Mental Test Score is applied.

Exclusion Criteria:

* Having serious vision and hearing loss,
* Having an orthopedic, vestibular, neurological or mental problem such as upper and lower extremity pathology that may prevent or limit the application of the test protocol,
* Having a diagnosis of postural hypotension,
* Lack of cooperation,
* Being in the recovery period of an acute disease was determined as an exclusion criterion.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The required sample size for validation studies was reported as 2-20 participants per item on the scale (14). HRERS consists of five questions, thus we included at least fifty participants. A total of 51 consecutive participants, inpatients of an orthopaedic clinic at university hospital, were recruited between 2021-2022 June.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Hopkins Rehabilitation Engagement Rating Scale-HRERS | 3-5 days (after every rehabilitatiom program)
  HRERS is a 5-item and practitioner completed scale used to rate behavioral observations of patients during acute inpatient rehabilitation.To evaluate the parameters of engagement in rehabilitation activities, the HRERS items rate the following: (I) the level of attendance at therapy sessions, (II) the attitude expressed by the patient toward his/her therapy, (III) the need for verbal or physical prompts to facilitate initiation or maintenance of engagement within the therapy session, (IV) the patient's acknowledgment of the need for therapy and (V) the patient's level of active participation in the therapy. This questionnaire evaluates five items on a 6-level-likert scale from 1 (never) to 6 (always). Higher scores indicate higher engagement levels.

SECONDARY OUTCOMES:
Functional Independence Measurement-FIM | 3-5 days (after every rehabilitatiom program)
  The FIM instrument is the functional assessment measure. The FIM includes 18 items that measure functional independence in 6 subscales: self-care, sphincter control, mobility, locomotion, communication, and social cognition.Each item is rated on a seven-point scale that represents different gradations of independence and reflects the amount of assistance the patient requires to perform a specific activity. Independence is categorized and scored as complete independence, 7; modified independence, 6; requires supervision or setup, 5; requires minimal contact assistance, 4; requires moderate assistance, 3; requires maximal assistance, 2; and requires total assistance, 1. The sum of all 18 items comprises the patient's total FIM score, which ranges from 18 to 126
Barthel Index | 3-5 days (after every rehabilitatiom program)
  Based on observation, this practitioner-reported index measures patients' functional status across 10 domains: faecal incontinence, urinary incontinence, personal care (cleaning teeth, shaving), using the toilet, feeding, transfers (e.g. chair to bed), walking, dressing, climbing stairs, and bathing (or showering). Scoring of individual domains range between 0 and 15 (at 5-point intervals): domains vary in the number of intervals offered. The total score is used which ranges from 0 (no functioning) to 100 (independent functioning)
European Quality of Life-5 Dimensions Questionnaire-EQ-5D | 3-5 days (after every rehabilitatiom program)
  Quality of life was assessed in hospital using EQ-5D, which consists of two tools: EQ. 5D descriptive system and EQ. 5D-VAS. The EQ. 5D descriptive system is a questionnaire evaluating 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) from which a score ranging from 0 to 1 (maximum health status) is derived. The EQ. 5D-VAS is a visual analogue scale ranging from 0 to 100 (maximum health status) where patients has to indicate the level of health status

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha BAŞKURT, Prof. Dr., Principal Investigator — Suleyman Demirel University
Locations (1):
- Menekşe ŞAFAK, Merkez, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No